CLINICAL TRIAL: NCT06521476
Title: Impact of Acetazolamide on Central Sleep Apnea Patients Receiving Medication for Opioid Use Disorder
Brief Title: Acetazolamide in Central Sleep Apnea Patients Using Medication for Opioid Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanjay R Patel (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Sanjay R Patel, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY23100016; R01DA059465 (NIH)
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Central Sleep Apnea Comorbid With Opioid Use
Keywords: Acetazolamide; Opioid Use Disorder; Medication for opioid use disorder (MOUD); Methadone; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 1:1 fashion to one of two parallel arms (active drug versus placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo pill matched to look like active drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Experimental): All participants in this group will receive one acetazolamide 250 mg pill in the evening for 7 days.
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): All participants in this group will receive one matching placebo pill in the evening for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Oral acetazolamide 250 mg daily for 7 days
  Arms: Acetazolamide
Drug: Placebo — Oral placebo daily for 7 days
  Arms: Placebo

SUMMARY:
Patients with opioid use disorder treated with either methadone or buprenorphine are at risk of developing central sleep apnea (CSA) from these medications. Investigators will conduct a mechanistic trial using acetazolamide, a medicine known to improve CSA in other settings, to determine if acetazolamide can improve CSA due to medication for opioid use disorder and whether this leads to physiologic changes that might lead to reduced drug craving. Patients treated with medication for opioid use disorder and who have central sleep apnea will be randomized to treatment with acetazolamide or matching placebo for 7 days. At the end of the 7 days, they will undergo an overnight sleep study to assess the impact on breathing during sleep as well as sleep quality. In addition, measures of sympathetic tone, anxiety, arousal, cognition, and drug craving will be measured to determine if treatment of CSA with acetazolamide can produce physiologic changes that might contribute to improved health.

DETAILED DESCRIPTION:
Medications used to treat opioid use disorder (MOUD) such as methadone and buprenorphine have been found to cause central sleep apnea (CSA), but the clinical ramifications are unclear. It has been hypothesized that the sleep fragmentation and intermittent hypoxemia caused by CSA from MOUD may lead to sympathetic activation, nocturnal arousal, increased anxiety, and cognitive impairment that may in turn increase drug craving and drug relapse. This mechanistic study will evaluate the potential adverse effect of CSA in patients on MOUD by evaluating the impact of acetazolamide to improve CSA and thereby lead to downstream physiologic changes in measures of sleep quality, sympathetic tone, nocturnal arousal, anxiety, cognitive functioning, and drug craving.

Eligible individuals will undergo an overnight research visit including overnight polysomnography, assessments of autonomic tone, sleep quality, nocturnal arousal, emotional distress, cognitive testing, and drug craving. Individuals with opioid-induced CSA will be randomized into a parallel-arm trial of acetazolamide vs. placebo with overnight research visit for outcome assessment at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients on Medication for Opioid Use Disorder (MOUD) with central sleep apnea.

Exclusion Criteria:

* Sleep-related Hypoventilation.
* Other causes of Central Sleep Apnea besides Opioid Use.
* Pregnancy.
* Contraindications for Acetazolamide.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Central Apnea Index (CAI) | 7 days
  The number of central apneas per hour of sleep, assessed by overnight polysomnography.
  * It can range from 0 to undefined events per hour.
  * Higher values indicate more severe central sleep apnea.

SECONDARY OUTCOMES:
Low frequency / high-frequency ratio (LF/HF ratio) | 7 days
  The ratio of low frequency to high frequency spectral power from heart rate variability analysis of electrocardiogram (ECG) collected during non-rapid eye movement (NREM) sleep on overnight polysomnography
Apnea Hypopnea Index (AHI) | 7 days
  The number of apneas plus hypopneas per hour of sleep on overnight polysomnography
  * It can range from 0 to undefined events per hour.
  * Higher values indicates severity of apneas and hypopneas.

OTHER OUTCOMES:
Overnight urinary norepinephrine levels | 7 days
  Overnight urinary norepinephrine concentration normalized to urinary creatinine concentration
Pre-ejection period | 7 days
  Pre-ejection period assessed by impedance cardiography
Pre-sleep Arousal Scale (PSAS) score | 7 days
  16-item questionnaire assessing level of nocturnal arousal
  * It can range from 16 to 80.
  * Higher scores indicate higher levels of nocturnal arousal.
Arousal Index | 7 days
  The number of cortical arousals per hour of sleep on overnight polysomnography.
  * It can range from 0 to undefined events per hour.
  * Higher values indicate more severe sleep disturbance.
Generalized Anxiety Disorder 7 (GAD-7) score | 7 days
  7-item questionnaire assessing anxiety symptoms
  * It can range from 0 to 21.
  * Higher scores indicate more severe anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance score | 7 days
  t-score derived from 8-item PROMIS sleep disturbance questionnaire
  * Population mean is 50 and standard deviation is 10.
  * Higher values indicate greater levels of sleep disturbance.
Opioid cue-induced drug craving | 7 days
  The mean craving score reported after exposure to visual opioid cues relative to craving scores after viewing neutral cues.
  * Mean craving score ranges from 0 to 10.
  * Higher scores indicate higher level of drug craving.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay R Patel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) from this clinical trial will be shared with other researchers. The IPD to be shared includes final closed dataset (after de-identification). All data will be released according to the specific timelines stated in the National Institutes of Health (NIH) Policy, ensuring no compromise to privacy, confidentiality, proprietary interests, national security, or law enforcement activities. These data will be submitted to a NIH-funded data registry for data sharing purposes.
Supporting Information: Study Protocol
Time Frame: The IPD will become available within 1 year of analysis of primary outcome. This data will be accessible on an NIH-sponsored platform for as long as the agency maintains it.
Access Criteria: IPD will be available through a NIH funded registry. Access to the IPD will be governed by the policies and procedures of NIH.